CLINICAL TRIAL: NCT04623515
Title: Exploring the Impact of Radiation Therapy on Pelvic Floor Disorders in Women Treated for Colorectal Cancer (RadPFD)
Brief Title: Radiation Therapy on Pelvic Floor Disorders in Women
Acronym: RadPFD
Status: Terminated | Type: Observational
Why Stopped: IRB closure, slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00069825; WFBCCC 01620 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
Keywords: Survivors of colorectal cancer; Lower bowel tract symptoms; Urinary incontinence; Irritative voiding symptoms; Voiding dysfunction; Bowel incontinence; Defecatory dysfunction; Lower urinary tract symptoms
MeSH Terms: conditions — Colorectal Neoplasms; Urinary Incontinence; Fecal Incontinence; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery Only Group: Participants will complete a questionnaires regarding demographics and medical history on a secured REDCap link.
  Interventions: Other: REDCap Questionnaires
- Surgery and Radiation Therapy Group: Participants will complete a questionnaires regarding demographics and medical history on a secured REDCap link.
  Interventions: Other: REDCap Questionnaires

INTERVENTIONS:
Other: REDCap Questionnaires — Once consent is obtained, the participants will be routed to a REDCap secure link. Participants will complete a questionnaires regarding demographics and medical history. Participants will also complete validated questionnaires regarding their lower urinary and bowel tract function and sexual health- International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ-FLUTS), Modified Manchester Health Questionnaire (MMHQ), PROMIS® v2.0 Brief Profile Sexual Function and Satisfaction (Female) and SF-12 ® .

SUMMARY:
Investigators propose a retrospective cohort study to examine the impact of radiation therapy on the global pelvic floor function of women who have completed the immediate surveillance period for colorectal cancer

DETAILED DESCRIPTION:
Primary Objective: To characterize the impact of radiation therapy on the lower urinary and bowel tract symptoms, (featuring urinary incontinence, irritative voiding symptoms, voiding dysfunction, bowel incontinence, and defecatory dysfunction) of female survivors of colorectal cancer 2-5 years after treatment.

Secondary Objectives:

* To characterize sexual dysfunctions present in female colorectal cancer survivors 2-5 years after treatment and to determine the impact of radiation therapy compared to surgical treatment alone.
* To examine the impact of radiation therapy on the sexual function of the partner of female survivors of colorectal cancer treated with radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Living, female patients.
* Age 18 or older with a diagnosis of colorectal cancer (current or past, regardless of Stage)-confirmed by pathology report - made between the years of 2015 and 2018.
* History of treatment for colorectal cancer in the Wake Forest Baptist Health System.
* Sexual partners of the above participants (subjects can participate even if they are not sexually active or if no sexual partner is available).
* English speaking.

Exclusion Criteria:

* No internet access.
* Non-English speakers (validated instruments are only available in English).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female survivors of colorectal cancer and their partners.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Urinary Dysfunction - International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) | Up to 4 months
  The ICIQ-FLUTS is a 12-item validated, self-administered questionnaire that is derived from the Bristol Female Lower Urinary Tract Symptoms (BF-LUTS) questionnaire and designed for use in women and to assess urinary symptoms and effects on quality of life. There are 3 subscales within this instrument to assess incontinence, voiding and filling. Investigators will specifically use the incontinence subscale as the primary outcome. The instrument is based on 5 questions, with possible answers on a 5-point scale (ranging from "never" to "all of the time"). Scoring is 0-48 with higher scores equaling to a greater bother with urinary dysfunction in participants.

SECONDARY OUTCOMES:
PROMIS® Brief Profile Sexual Function and Satisfaction (Female) | Up to 4 months
  This is a 14-item validated questionnaire that has been validated for use in cancer populations to assess female sexual function. Scoring is 0-100 with lower numbers indicating worse sexual function.
Bowel Dysfunction - Modified Manchester Health Questionnaire | Up to 4 months
  This is a 31-item patient reported outcome measure that is designed to assess degree and severity of bowel dysfunction and the impact of this dysfunction on quality of life. Scoring is 0-100 with higher scores indicating worse bowel function.
PROMIS® Brief Profile Sexual Function and Satisfaction- Male or Female Partners | Up to 4 months
  The PROMIS® Brief Profile Sexual Function and Satisfaction is an 11-item validated questionnaire that has been validated in a heterogeneous population to assess partner sexual function. Scoring is 0-100 with lower numbers indicating worse sexual function.
Dyadic Adjustment Scale-Short Form (DAS-7) Questionnaire - Couple Relationship | Up to 4 months
  This is a 7-item questionnaire to assess the quality of dyadic relationship designed for cohabitating or married couples. Score range is 0-36 with higher scores indicating better function.
Short Form-12 Questionnaire - General Health and Well Being | Up to 4 months
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. Scoring is 0-100 with higher scores indicating better function in the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Candace Parker-Autry, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No